CLINICAL TRIAL: NCT03479710
Title: Fecal Microbiota Transplantation for Eradication of Intestinal Colonization of Carbapenem-resistant Enterobacteriaceae and Vancomycin-resistant Enterococcus: a Pilot Study
Brief Title: Fecal Microbiota Transplantation for CRE/VRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT protocol v.2 10Oct2017
Record Dates: First submitted 2018-01-23; First posted 2018-03-27 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Antimicrobial Resistance; Colonization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT infusion (Experimental): FMT will be performed using frozen donor stool samples obtained from the stool bank of CUHK. 100-200ml of FMT solution or sterile saline will be infused over 2-3 minutes into the distal duodenum or jejunum via OGD.
  Interventions: Biological: FMT infusion
- Control (No Intervention): No FMT infusion.

INTERVENTIONS:
Biological: FMT infusion — Fecal microbiota transplantation via OGD
  Arms: FMT infusion

SUMMARY:
Multidrug-resistant organisms (MDRO) present an increasingly serious public health threat to the global community.The prevalence of various MDRO, including carbapenem-resistant Enterobacteriaceae (CRE) and vancomycin-resistant Enterococcus (VRE), has been increasing worldwide, and some have become endemic in certain countries. Data from the Hospital Authority showed that the number of carbapenemase- producing Enterobacteriaceae (CPE) cases increased from 36 in 2012 to 134 in 2015. A large outbreak of VRE involving >200 patients was recently reported in a tertiary hospital in Hong Kong.

The primary site of colonization and persistence of most MDRO is in the gastrointestinal tract. Carriage can persist for months, with up to 40% of individuals still having colonization one year after hospital discharge. Outbreaks of MDRO have been reported in hospitals and long-term care facilities. Around 10% of patients colonized with MDRO would develop clinical infections by the same organism. Infections caused by these MDRO carry significant morbidity and high mortality of up to 50%, however, there is no proven therapy for eradication of intestinal colonization of MDRO.

There is accumulating evidence showing that the gut microbiota plays an important role in the control of intestinal colonization and infection by pathogenic bacteria. Administration of obligate anaerobic commensal bacteria to mice has been shown to markedly reduce VRE colonization. Preliminary evidence, mainly from anecdotal reports, have shown that fecal microbiota transplantation (FMT) in human carriers of MDRO were safe and potentially effective in eliminating intestinal colonization by various MDRO, including CRE and VRE, even in immunocompromised patients. Therefore, investigators hypothesize that FMT will be safe and potentially effective in eradicating intestinal colonization of CRE and VRE.

This is a prospective pilot study to evaluate whether FMT is safe and effective to eradicate intestinal colonization of CRE and VRE.

ELIGIBILITY:
Inclusion Criteria:

For cases:

1. Age ≥18 years old
2. Two or more stool or rectal swab positive for CRE or VRE at least one week apart.

   [CRE is defined as presence of any Enterobacteriaceae with resistance to any of the carbapenems. VRE is defined as presence of Enterococcus species resistant to vancomycin.]
3. Not receiving antimicrobial therapy for at least 48 hours prior to infusion of FMT

For controls:

1. Age ≥18 years old
2. Two or more stool or rectal swab positive for CRE or VRE at least one week apart.
3. Not receiving antimicrobial therapy for at least 48 hours prior to infusion of FMT
4. Refuse to consent for FMT infusion but consent for other study procedures listed in the protocol.

Exclusion Criteria:

1. Active infection with CRE or VRE requiring antimicrobial therapy
2. Pregnancy
3. Active gastrointestinal tract infection or inflammatory disorders
4. Recent intra-abdominal surgery
5. Short gut syndrome
6. Use of medications which alter gastrointestinal motility at the time of inclusion
7. Post-allogeneic hematopoietic stem cell transplant patients with history of gastrointestinal tract graft versus host disease
8. Presence of intra-abdominal device which would increase risk of peritonitis
9. ANC <500/mm3
10. HIV infection with CD4 <200 cells/mm3
11. On chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Intestinal colonization of CRE/VRE | 2 weeks to 12 months
  Absence of intestinal colonization of CRE/VRE

SECONDARY OUTCOMES:
Adverse events | 12 months post FMT
  Incidence, severity and relatedness of adverse events
Intestinal microbiota | Before and 12 months after FMT
  Changes in intestinal microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lui, Principal Investigator — CUHK
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided